CLINICAL TRIAL: NCT05313438
Title: Cardiac Pulmonary Nerve STIMulation in Acute Decompensated Heart Failure
Brief Title: The STIM-ADHF Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardionomic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-1108-001
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Neurostimulation; Contractility; Right Pulmonary Artery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CPNS Therapy (Experimental): Endovascular stimulation of the cardiac autonomic nerves in addition to standard of care.
  Interventions: Device: CPNS Therapy

INTERVENTIONS:
Device: CPNS Therapy — Endovascular stimulation of the cardiac autonomic nerves in addition to standard of care

SUMMARY:
The STIM-ADHF Study is a multi-center, observational study to assess the performance and safety of the CPNS System in patients with ADHF.

DETAILED DESCRIPTION:
The CPNS System is a neuromodulation system used to treat ADHF, a sudden or slow deterioration of chronic heart failure. The CPNS system is intended to provide acute (≤ 5 days) endovascular stimulation of the cardiac autonomic nerves in the right pulmonary artery (PA) in hospitalized ADHF patients. The system consists of an acute temporary neuromodulation stimulation catheter placed in the right pulmonary artery via venous access and a custom stimulator, denoiser, and associated cables. The CN2 Catheter is delivered to the right PA and provides an inotropic and/or lusitropic therapeutic effect by electrical stimulation to the terminal sympathetic nerve branches within the cardio-pulmonary plexus. The study will be conducted at up to 20 study sites worldwide. Up to 50 subjects who meet the eligibility criteria, will be enrolled, treated in-hospital with the Cardionomic CPNS System, monitored closely throughout the hospitalization and followed through 30 days post hospital discharge to evaluate the effect of the CPNS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital or planned to be admitted with a principal diagnosis of acute decompensated heart failure
* BMI adjusted BNP ≥ 500 pg/mL or NT-proBNP ≥ 2000 pg/mL
* LVEF ≤ 50%
* At least one sign/symptom of fluid overload
* At least one of the following:
* Inadequate diuretic response
* At least one sign or symptom of low perfusion

Exclusion Criteria:

* Received an inotrope during current hospitalization
* Requires mechanical support
* Cardiogenic shock or impending cardiogenic shock
* Multi-organ failure
* Systolic blood pressure < 80mmHg or > 140mmHg
* Symptomatic hypotension
* eGFR < 25 mL/min/1.732
* Severe hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of related adverse events | Enrolment to 30 Days post hospital discharge
  The following measures will be characterized in all enrolled subjects: occurrence of all procedure, device and therapy related adverse events, serious adverse events and deaths

CONTACTS AND LOCATIONS:
Locations (6):
- Hungary (3):
  - Semmelweis University, Heart and Vascular Center, Budapest
  - Hearth Faculty of Medicine, University of Pécs, Pécs
  - Szegedi Tudományegyetem ÁOK, Szeged
- American Heart of Poland, Bielsko-Biala, Poland
- Slovakia (2):
  - Stredoslovenský Ústav srdcových a Cievnych Chorȏb, a.s., Banská Bystrica
  - CINRE s.r.o, Bratislava